CLINICAL TRIAL: NCT06319976
Title: Effect of Rotator Cuff Training on Hand Grip Strength and Endurance in Adults With Different Body Mass Index
Brief Title: Effect of Rotator Cuff Training on Hand Grip in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Atef Mohammed Mohammed, Principal investigator at department of basic science , Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004883
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Hand Grasp
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open chain exercises for rotator cuff muscles and advices for postural correction (Experimental): Group will be subdivided into three subgroups according to their body mass index to normal, over weight and obese type1. All subjects will receive open chain exercises for rotator cuff muscles and advices for postural correction.
  Interventions: Other: open chain exercises for rotator cuff muscles; Other: Advices for postural correction
- Advices for Postural correction (Active Comparator): Group will be subdivided into three subgroups according to their body mass index to normal, over weight and obese type1. All subjects will receive advices for postural correction. .
  Interventions: Other: Advices for postural correction

INTERVENTIONS:
Other: open chain exercises for rotator cuff muscles — open chain exercises for rotator cuff muscles, three times per week for six weeks.
  Arms: open chain exercises for rotator cuff muscles and advices for postural correction
Other: Advices for postural correction — Advices for postural correction like neutral position of head and neck, aliening the shoulder and hip and using a foot stool to rest the feet.

SUMMARY:
Purpose of the study:

* To investigate the effect of rotator cuff training on hand grip strength in adults with different body mass index.
* To investigate the effect of rotator cuff training on hand grip static endurance in adults with different body mass index.
* To investigate the effect of rotator cuff training on hand grip dynamic endurance in adults with different body mass index.
* To investigate the effect of rotator cuff training on upper limb function in adults with different body mass index.

DETAILED DESCRIPTION:
Rotator cuff muscles are considered to be the key dynamic muscles in shoulder stabilization since they contribute significantly to shoulder stability in a number of different ways. They work not only as a dynamic stabilizer but also as static stabilizers because of their orientation and location around the shoulder joint. Several studies revealed the strong relationship between the rotator cuff muscles and hand grip strength. Studies proved the strong correlation between grip strength and rotator cuff strength ,which suggests that assessment of grip strength could be used to monitor the function of the rotator cuff, once baseline readings have been attained during training and rehabilitation .

Previous publications revealed significant positive associations between handgrip strength, body mass index (BMI) and physical activity in adult men and women. Worldwide, 31.1% of adults are reported to be physically inactive. Some studies and reports indicate that 20% of the global populace within the age range of 18-64 years comply with the minimum physical activity guidelines for improved health. Overweight and obesity are identified as a constant negative influence on physical activity, regardless of age.

Studies proved that weight, height, and BMI have a significant correlation on hand grip strength. As the weight increase hand muscle strength and endurance time also decrease.

Subjects in this study will be recruited from the students , employees and faculty members of the faculty of physical therapy, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Subjects of both genders their ages between (18 : 35) years old.
2. Body mass index between (18.5 : 34.9 ) Kg/ m2.
3. Dominant hand is the right hand.

Exclusion Criteria:

The subjects will be excluded if they have:

1. Traumatic conditions of the upper limb.
2. Previous orthopedic disorders or neurological deficit of the upper limb.
3. Previous surgery of the upper limbs.
4. Any sensory problems.
5. Neuromuscular disease like multiple sclerosis.
6. Pregnancy.
7. Cancer Patients.
8. Subjects under chemotherapy.
9. Immunodeficiency diseases.
10. Psychological disorders (depression - anxiety).
11. Chronic diseases as (diabetes - hypertension).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength | up to six weeks
  The JAMAR Hydraulic hand dynamometer is used to measure hand grip strength in (Kg) , It will be evaluated before and after training for each subject in both groups. Each subjects will be asked to grasp the handle with the dominant hand and perform hand grip with maximum effort only during exhalation and after a verbal cue given by the examiner " one, two, three, go". The subjects will be instructed to maintain maximum contraction for 5 seconds. Three measurements will be taken with a rest interval of 60 seconds between trials in order to avoid muscle fatigue during the assessment and the average of the three measurements will be calculated to measure hand grip strength.

SECONDARY OUTCOMES:
Hand grip static endurance | up to six weeks
  It will be evaluated before and after training for each subject in both groups by using JAMAR Hydraulic hand grip dynamometer, Subjects will be seated in initial position. They will be asked to grip the hand grip dynamometer at 60% of their maximum voluntary contraction (MVC). The duration for which they maintained the grip strength will be noted in seconds. Subjects will be verbally encouraged to maintain the contraction at the set target for as long as possible. The test will be terminated when the subjects fail to maintain the 60% MVC for two consecutive times. Two recordings will be obtained with a gap of five minutes between each effort.
Hand grip dynamic endurance | up to six weeks
  It will be evaluated before and after training for each subject in both groups by using JAMAR Hydraulic hand dynamometer, After static hand grip endurance test, the subjects will perform the dynamic hand grip endurance test. Subjects will be instructed to give repetitive contractions at 60% of their maximal voluntary contraction (MVC) on the beat of the metronome set at 70 beeps per minute until fatigue set in and they will be no longer able to produce the same intensity of contraction. Number of repetitions will be measured.
Upper limb function | up to six weeks
  Each subject in both groups will receive and fill the items of Arabic version of The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire before and after training. The DASH is a 30-item self-report questionnaire designed to evaluate impairments and activity limitations, as well as participation restrictions for both leisure activities and work. Response options range from 1 to 5 (1: no difficulty; 2: mild difficulty; 3: moderate difficulty; 4: severe difficulty; 5: unable). The DASH produces scores between 0 and 100 for each module, in which a high DASH score indicates severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Saleh, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol